CLINICAL TRIAL: NCT00905983
Title: Phase II Study of Biweekly Gemcitabine and Docetaxel as First Line Treatment for Advanced Disease in Elderly Non Small Cell Lung Cancer (NSCLC) Patients.
Brief Title: Biweekly Gemcitabine and Docetaxel as First Line Treatment for Advanced Disease in Elderly Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Vicente Alberola Candel, ASOCIACIÓN TERAPEUTICA EN HEMATOLOGÍA Y ONCOLOGÍA MÉDICAS H. ARNAU DE VILANOVA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPNM-ANC-07
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell; Elderly patients; Docetaxel; Gemcitabine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine and Docetaxel (Experimental): Patients received biweekly docetaxel 50 mg/m2 iv, Gemcitabine 2000 mg/m2 iv days 1 and 14.
  Interventions: Drug: Gemcitabine and Docetaxel

INTERVENTIONS:
Drug: Gemcitabine and Docetaxel — Docetaxel 50 mg/m2, IV, and Gemcitabine 2000 mg/m2, IV, on day 1 and 14 of each 28 day cycle. Number of Cycles: 6

SUMMARY:
Lung cancer is one of the most common malignancies worldwide and the leading cause of cancer-related deaths in Western countries. Standard treatment for patients with good performance status (PS) stage IIIB/IV NSCLC currently includes a two-drug platinum-based chemotherapy regimen, but optimum treatment for elderly patients is less well-defined due to platinum related toxicities. Several drugs with novel mechanisms of action and significant activity in NSCLC have been developed; including docetaxel and gemcitabine that are also active in patients previously treated with cisplatin-based regimens and have a more favorable toxicity profile. The more favorable toxicity profile of docetaxel and gemcitabine supports its use as first-line chemotherapy, especially in patients with severe comorbidities as elderly patients. To improve the therapeutic index of this combination, the investigators performed a study with biweekly gemcitabine and docetaxel in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced NSCLC.
* Stage III with pleural effusion and stage IV.
* Patients are 70 years old.
* Patients with 1 > ECOG PS =1.
* Patients must have at least one measurable lesion, no previously irradiated.
* Life expectancy of at least 12 weeks.
* Adequate organ function according to the following criteria:

  * Bone marrow: ANC >= 2.0x10(9)cells/L; Platelet count >= 100x10(9)cells/L; Leukocyte count >= 4000x10(6)/L; Hemoglobin >= 10 g/dL.
  * Liver function: Bilirubin <= 1.5 X ULN; Alkaline phosphatase <= 5 x ULN;AST and ALT <= 1.5 x ULN.
  * Renal function: serum creatinine <= 2mg/dL.

Exclusion Criteria:

* Prior systemic chemotherapy for advanced disease.
* Patients with symptomatic brain metastases.
* No measurable bone metastases or malignant pleural effusion as only measurable lesion.
* History of prior malignancies, except curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years.
* History of hypersensitivity reaction to study drugs.
* Concurrent treatment with other experimental drugs.
* Current peripheral neuropathy NCI grade 2.
* Participation in clinical trials within 30 days of study entry.
* Major surgery, open biopsy or traumatic lesion 28 days before to study start.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate = sum of complete and partial tumour responses divided by the number of included patients | 2 & 4 months

SECONDARY OUTCOMES:
Overall survival | time from study entry to death from any cause
Toxicity | biweekly
Duration of response | time from first response (CR or PR) to tumor progression
Time to progression | time from study entry to observed tumor progression or death due to progression disease
Measurement of quality of life | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Juan, Doctor, Study Director — Hospital Arnau de Vilanova de Valencia; Alfredo Sánchez, Doctor, Principal Investigator — Hospital Provincial de Castellón; José Muñoz, Doctor, Principal Investigator — H. Universitario Dr. Peset; Sonia Maciá, Doctor, Principal Investigator — Hospital General de Elda; Vicente Giner, Doctor, Principal Investigator — Hospital de Sagunto; José Gómez, Doctor, Principal Investigator — Hospital Universitario La Fe; Gaspar Esquerdo, Doctor, Principal Investigator — Hospital Clínica de Benidorm; Antonio López, Doctor, Principal Investigator — Hospital San Juan de Alicante; Francisco Aparisi, Doctor, Principal Investigator — Hospital Virgen de los Lirios; Miguel A. Muñoz, Doctor, Principal Investigator — Instituto Valenciano de Oncología; Silvia Catot, Doctor, Principal Investigator — Hospital Althaia, Xarxa Asistencial de Manresa
Locations (11):
- Spain (11):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital San Juan de Alicante, Alicante, Alicante
  - Hospital Clínica de Benidorm, Benidorm, Alicante
  - Hospital General de Elda, Elda, Alicante
  - Hospital Althaia, Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia